CLINICAL TRIAL: NCT05292638
Title: A Randomized, Double-blind, Active-controlled, Single-center Phase I Trial to Investigate the Safety and Efficacy of CKDB-501A in Subjects With Moderate-to-severe Glabellar Lines
Brief Title: Safety and Efficacy of CKDB-501A in Subjects With Moderate-to-severe Glabellar Lines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CKD Bio Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CKDB-BAGL-101
Record Dates: First submitted 2022-02-23; First posted 2022-03-23 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Glabellar Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: Active-controlled
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CKDB-501A (Experimental)
  Interventions: Drug: CKDB-501A
- Botox® (Active Comparator)
  Interventions: Drug: Botox®

INTERVENTIONS:
Drug: CKDB-501A — Intramuscular injection CKDB-501A
  Arms: CKDB-501A
Drug: Botox® — Intramuscular injection Botox®
  Arms: Botox®

SUMMARY:
A single-center, randomized, double-blind, single-injection, active-controlled, parallel-design study to evaluate the safety and efficacy of CKDB-501A in Glabellar lines.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with at least moderate glabellar frown lines at maximum frown using the severity score of at least 2(moderate) on the Facial Wrinkle Scale (4-point FWS)

Exclusion Criteria:

* Any medical condition (e.g., myasthenia gravis, Lambert-Easton syndrome, amyotrophic lateral sclerosis, etc.) that can affect the neuromuscular function
* History of facial nerve paralysis or ptosis
* Significant facial asymmetry
* Subjects with skin abnormalities such as infection, dermatologic disorders, scars, etc. at potential injection sites
* Previous treatment with any serotype of botulinum toxin products within 24 weeks (6 months) prior to Screening or planning to receive treatment with botulinum toxin during the study period
* Previous treatment with retinoids (isotretinoin, alitretinoin, etc.)

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events | up to week 12
  severity and frequency of reported adverse events

SECONDARY OUTCOMES:
Proportion of subjects with improvement in investigator-assessed glabellar line severity at maximum frown at each follow-up visit | Week 4, 8, 12
  using the 4-point FWS (Facial Wrinkle Scale, range from 0(None) to 3(Severe))
Proportion of subjects with improvement in investigator-assessed glabellar line severity at rest at each follow-up visit | Week 4, 8, 12
  using the 4-point FWS (Facial Wrinkle Scale, range from 0(None) to 3(Severe))
Changes in the investigator-assessed glabellar line severity score from baseline at each follow-up visit | Week 4, 8, 12
  using the 4-point FWS (Facial Wrinkle Scale, range from 0(None) to 3(Severe))
Proportion of subjects with improvement in subject's assessment of glabellar line severity at each follow-up visit | Week 4, 8, 12
  using the Subject Assessment 9-grade Scale(range from -4(very marked worsening) to +4(complete inprovement)
Subject-assessed satisfaction scale at each follow-up visit | Week 4, 8, 12
  using the Subject Satisfaction 7-point Scale(range from 1(very dissatisfied) to 7 (very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: beomjoon Kim, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (1):
- Chung-Ang University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No